CLINICAL TRIAL: NCT01958203
Title: Venous Thromboembolism Prophylaxis in a Tertiary UAE Hospital: Comparison of Clinical Practice Guidelines.
Acronym: VTE
Status: Completed | Type: Observational
Sponsor: Ministry of Health, United Arab Emirates (Other Government)
Responsible Party: Principal Investigator, Dr. Ghada Al Tajir, Director of Clinical Research Centre, Ministry of Health, United Arab Emirates
Other Study IDs: 122012-11
Record Dates: First submitted 2013-09-29; First posted 2013-10-09 (Estimated); Last update posted 2013-10-09 (Estimated); Status verified 2013-10

CONDITIONS: Venous Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
Study Title:Assessment of Adherence to Guidelines for Thromboprophylaxis in a Tertiary United Arab Emirates (UAE) hospital

Study Site: Al Qassimi Hospital, United Arab Emirates

Study Objectives:

The primary objective of this study is assessment of appropriateness of VTE prophylaxis administered to critically ill and surgical patients for whom pharmacologic treatment is indicated according to the American College of Chest Physicians (ACCP) 2012 guidelines.

The secondary objective is to:

1.Identify some causes of inadequate VTE prophylaxis in different patient populations, such as prescribing problems and errors at the level of administration.

Study Design: Cross sectional retrospective observational study

Sample size: Approximately 400

Study Population:

Inclusion criteria

Patients who meet the following criteria will be included:

1. Patients aged 18 and above.
2. Patients admitted to any of the critical care units, or the general or orthopaedic surgical wards.
3. Patients who have been in hospital more than 24 hours.
4. Caprini score > 1 (see procedure)

Exclusion criteria

Patients with any of the following criteria will be excluded:

1. Patients who have been admitted to a critical care unit and transferred out to a non surgical unit within 24 hours of admission.
2. Patients receiving oral anticoagulant therapy for indications other than VTE prophylaxis or treatment, such as atrial fibrillation and prosthetic heart valves.

Study Outcome Measurements:

The main outcome measure of interest is to determine the proportion of patients who have received inappropriate or inadequate VTE prophylaxis considering their calculated risk factor compared to the recommended prophylactic measures for that risk.

Secondary outcome measures are to identify whether there is inadequate VTE prophylaxis because of medication errors such as missed doses or wrong doses given.

Study Duration: 4 months

Statistical Analysis Data was entered into Microsoft Excel® and subsequently checked to ensure accurate data entry and correct any errors. It was subsequently exported into SPSS version 20 where it will be analysed.Quantitative data such as age was expressed mean (± standard deviation). Categorical data such as gender, risk factors for bleeding, type of mechanical and pharmacologic prophylaxis, missed doses and wrong doses were expressed as number and percentage of population.The student's t-test was used to analyse parametric data. The Pearson Chi-Square Test and Wilcoxon Rank sum test were used to analyse non parametric data. Simple and multiple logistic regression analysis was done to identify factors that are associated with inappropriate VTE prophylaxis. Factors that were included in the analysis included: age, type of admission (medical or surgical), area of admission (critical care, general surgery, orthopaedic surgery), Caprini score, and inappropriate VTE prophylaxis as the outcome. A p-value of less than 0.05 was be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 and above.
2. Patients admitted to any of the critical care units, or the general or orthopaedic surgical wards.
3. Patients who have been in hospital more than 24 hours.
4. Caprini score > 1 (see procedure)

Exclusion Criteria:

1. Patients who have been admitted to a critical care unit and transferred out to a non surgical unit within 24 hours of admission.
2. Patients receiving oral anticoagulant therapy for indications other than VTE prophylaxis or treatment, such as atrial fibrillation and prosthetic heart valves.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The targe sample is paients in critical care wards and orthopaedic surgery patients. All patients will be screened at discharge. Those who fulfill the inclusion/exclusion criteria will go on to have a thromboembolism risk assessment using the CapriniRisk Assessment Model. Those who have a score > 1 will be included for assessment of their VTE prophylaxis (from medical records). Approximately 60 patients are admitted into critical care units and 40 general and orthopaedic surgical patients are admitted to the surgical wards per month, giving a total sample of around 400 patients.
Sampling Method: Non-Probability Sample
Enrollment: 386 (Actual)
Dates: Start 2013-01; Primary Completion 2013-08 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Number of patients receiving inappropriate or inadequate VTE prophylaxis | 2 weeks
  Case Report Form Analysis Form

SECONDARY OUTCOMES:
Number of patients receiving inadequate VTE prophylaxis due to medication errors, missed doses etc. | 2 weeks
  Case Report Form Analysis Form

CONTACTS AND LOCATIONS:
Overall Officials: Ghada Al Tajir, Ph.D, Principal Investigator — Clinical Research Centre, Ministry of Health, United Arab Emirates